CLINICAL TRIAL: NCT01427816
Title: A Randomized, Double Blind, Placebo Controlled, Phase II Study of KCT-0809 in Patients With Dry Eye Syndrome
Brief Title: A Phase II Study of KCT-0809 in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCT1202
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- KCT-0809 ophthalmic solution, low dose (Experimental)
  Interventions: Drug: KCT-0809
- KCT-0809 ophthalmic solution, high dose (Experimental)
  Interventions: Drug: KCT-0809
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KCT-0809
  Arms: KCT-0809 ophthalmic solution, low dose
Drug: KCT-0809
  Arms: KCT-0809 ophthalmic solution, high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of KCT-0809 compared to placebo in patients with dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Corneal and conjunctival damage
* Insufficiency of lacrimal secretion
* Ocular symptom

Exclusion Criteria:

* Severe ophthalmic disorder
* Punctual plugs or surgery for occlusion of the lacrimal puncta

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180

PRIMARY OUTCOMES:
Corneal staining score | 6 weeks

SECONDARY OUTCOMES:
Conjunctival staining score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsumi Hontani, Study Director — Clinical Development Department, Kissei pharmaceutical Co., Ltd.
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan